CLINICAL TRIAL: NCT03043586
Title: Treatment Patterns and Treatment Outcomes in a New York City Based Cohort of 520 Patients With Acromegaly
Brief Title: Treatment Patterns and Treatment Outcomes for Acromegaly
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Principal Investigator, Pamela U. Freda, Professor of Medicine, Columbia University
Other Study IDs: AAAQ6709
Record Dates: First submitted 2017-01-30; First posted 2017-02-06 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Acromegaly
Keywords: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood will be sampled for fasting measurements of growth hormone (GH) and insulin Growth Factor 1 (IGF-1) and patients will undergo an oral glucose tolerance test (OGTT) with blood drawn before and 60, 90 and 120 minutes after a 75 g. dextrose drink.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment Pattern: The first phase of this study will be to contact all subjects in the cohort by a mailing introducing them to the study. This will be followed by a phone call and administration of a questionnaire by phone or by mail. A phone script will be utilized to obtain verbal informed consent from subjects for this phase of the study. The questionnaire will collect current information on acromegaly treatment, morbidities and other relevant history. Subjects will provide verbal consent to participate in this questionnaire part of the study and review of their medical records by the PI and study staff.

SUMMARY:
This is a human, prospective and retrospective, single-center study of patients who have undergone treatment for acromegaly in New York City since 1981. The project will characterize, among other factors, the treatment methods received by patients, who administered the treatments and the success of this therapy in terms of biochemical control.

DETAILED DESCRIPTION:
The first phase of this study will be to contact all subjects in the cohort by a mailing introducing them to the study. This will be followed by a phone call and administration of a questionnaire by phone or by mail. The questionnaire will collect current information on acromegaly treatment, morbidities other relevant history. Subjects will provide verbal consent to participate in this questionnaire part of the study and review of their medical records by the Principal Investigator (PI) and study staff.

In the second phase of the study, subjects will be invited to come for a visit that will be conducted by the PI and study staff at the Pituitary Center of Columbia University Irving Medical Center. At this visit written informed consent will be obtained. The investigators will review the subjects' medical history that is obtained from the subject and review any records and laboratory test results provided by the subject and conduct clinical and laboratory assessments. Although all subjects participating in Phase 1 will be invited to participate, it is estimated that 120 of the subjects invited will come for the one visit over the 2-year time frame of this study.

In the third phase of the study a chart review for collection will be conducted and all data will be compiled. All subjects agreeing to participate, both in person and by mail, a chart review of all relevant patient data including demographic, clinical, biochemical, surgical and follow up information. Data from questionnaires and record reviews will be compiled for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females.
* Ages 18 and over.
* Presenting to the PI or one of the sub-investigators for evaluation of acromegaly.
* Must be an Acromegaly subject that have undergone Pituitary surgery with Dr. Bruce or Dr. Post or Present it to principal investigator Dr. Pamela Freda at the Neuroendocrine Unit at Columbia University Medical Center for evaluation of Acromegaly.

Exclusion Criteria:

* Subjects who are unwilling to comply with the procedures outlined in the study.
* Subjects who do not have the ability to fully comprehend the nature of the study, to follow instructions, and/or cooperate with study procedures.
* Not being treated for acromegaly either by Dr. Bruce, Dr. Post or Dr. Freda.
* Are unwilling to provide informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population for this study is a cohort of 520 adult patients who have undergone treatment for acromegaly in NYC since 1981. The cohort is predetermined based on the patients who have previously undergone pituitary surgery for acromegaly with our two collaborating Neurosurgeons. Based on prior studies, the population has no gender predilection and no racial or ethnic predisposition and thus the ethnic mix of the cohort reflects the population of the NY metropolitan area that is referred to the study center.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients that have received surgery as first line therapy | At 5 years of therapy
  Frequency of each type of acromegaly therapy and rates of treatment by surgery alone, somatostatin analog, pegvisomant, radiotherapy and combinations of each of these therapies in the cohort will be recorded and determined. The expected result is that more than 90% of our cohort has received surgery as first line therapy and only a minority has received primary medical therapy.

SECONDARY OUTCOMES:
Number of patients with IGF-1 levels remaining elevated | At 5 years of therapy
  This is to identify patients who are not optimally managed since their IGF-1 levels remain elevated.
Hypertension Rate | At 5 years of therapy
  This is to identify if hypertension is affected by how treatment is managed.
Diabetes Mellitus Rate | At 5 years of therapy
  This is to identify if diabetes mellitus is affected by how treatment is managed.
Sleep Apnea Rate | At 5 years of therapy
  This is to identify if sleep apnea is affected by how treatment is managed.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela U Freda, MD, Principal Investigator — Columbia University
Locations (1):
- Neuroendocrine Unit at Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided